CLINICAL TRIAL: NCT01095042
Title: Etude de la réactivité émotionnelle Des Patients MICI ou SII
Brief Title: Cognition and Emotion in the SII and IBD
Acronym: EMOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: French National Society of Gastroenterology (Other); Association François Aupetit (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0817; 2008-A00994-51 (Registry Identifier: ID RCB)
Record Dates: First submitted 2010-02-22; First posted 2010-03-29 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Irritable Bowel Syndrome; Inflammatory Bowel Disease (IBD); Crohn's Disease(CD); Ulcerative Colitis
Keywords: HRV; emotion; cognition; stress; cortisol; Autonomic nervous system
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Experimental): 30 Asymptomatic Healthy Volunteers Intervention : Observation of emotional behavior in asymptomatic healthy volunteers subjected to stress.
  Interventions: Behavioral: emotion
- Experimental group (Experimental): Persons reached by digestive pathologies (SII or IBD). Group SII : 30 patients Group IBD: 60 patients (30 patients RCH and 30 patients CD)
  Intervention : Observation of emotional behavior in person affected by digestive pathologies subjected to stress.
  Interventions: Behavioral: emotion

INTERVENTIONS:
Behavioral: emotion — Show that the susceptibility in the stress (recording of Heart Rate Variability;viewing films;...) is more important at the person affected by digestive pathologies (SII or IBD) in forgiveness than to unhurt subjects of pathologies.
  Other Names: STRESS

SUMMARY:
The study aims at showing that the susceptibility in the stress is more raised at the person affected digestive pathologies (SII or IBD) in forgiveness than healthy subjects.

DETAILED DESCRIPTION:
The objective of the study which we wish to lead consists in looking for, at the patients SII and IBD in forgiveness, the existence of a correlation between the rate of cortisol(Hormone of the stress) and the level of HRV (Heart Rate Variability) to estimate the inhibitive fronto-amygdalien tonus.

So we make the hypothesis that the persons affected by digestive pathologies of type SII or IBD would present an emotional and physiological vulnerability more important than unhurt subjects of pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SII :Membership to the Social Security,SII defined according to the criteria Rome III.
* Patients with IBD :Membership to the Social Security,patients with a ulcerative colitis(UC) or a Crohn's disease (CD)ileal and/or colic.

Exclusion Criteria:

* Existence of a severe affectation on the general plan (cardiac,respiratory,hematological,renal,hepatic,cancerous),
* Subject diabetic,
* Pregnant or breast-feeding woman,
* Subject included in another clinical and\or therapeutic trial or having been included in a clinical and\or therapeutic trial for less than a month,
* Subject presenting a psychiatric pathology evident,
* Person under guardianship.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2008-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
RATE PLASMATIQUE OF CORTISOL COUPLED WITH THE CARDIAC VARIABILITY | 24 MONTHS

SECONDARY OUTCOMES:
SCORES OF DEPRESSIVE SYMPTOMATOLOGIE AND ANXIETY, RATE PLASMATIQUES OF CATECHOLAMINES, LEPTINE, ADIPONECTINE AND PRO-INFLAMMATORY CYTOKINES. | 24 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Bonaz, MD-PhD, Principal Investigator
Locations (1):
- Hôpital Michallon-CHU Grenoble, Grenoble, France

REFERENCES:
- [Background] Pellissier S, Dantzer C, Canini F, Mathieu N, Bonaz B. Psychological adjustment and autonomic disturbances in inflammatory bowel diseases and irritable bowel syndrome. Psychoneuroendocrinology. 2010 Jun;35(5):653-62. doi: 10.1016/j.psyneuen.2009.10.004. Epub 2009 Nov 11. PMID 19910123
- [Background] Graff LA, Walker JR, Clara I, Lix L, Miller N, Rogala L, Rawsthorne P, Bernstein CN. Stress coping, distress, and health perceptions in inflammatory bowel disease and community controls. Am J Gastroenterol. 2009 Dec;104(12):2959-69. doi: 10.1038/ajg.2009.529. Epub 2009 Sep 15. PMID 19755973
- [Background] Pellissier S, Dantzer C, Canini F, Mathieu N, Bonaz B. Toward a definition of a global psycho-physiological criterion of vulnerability to relapse in inflammatory bowel diseases. Am J Gastroenterol. 2010 Jun;105(6):1446-7. doi: 10.1038/ajg.2009.763. No abstract available. PMID 20523319